CLINICAL TRIAL: NCT04579549
Title: Repeat Saliva Testing for SARS-CoV-2 Using RT-LAMP Assay
Brief Title: Repeat Testing for SARS-CoV-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-1142; A536300 (Other: UW Madison); SMPH/PATHOL-LAB MED/ANAT PATH (Other: UW Madison); Protocol Version 8/17/2020 (Other: UW Madison); 5P51OD011106-59 (NIH)
Record Dates: First submitted 2020-10-06; First posted 2020-10-08 (Actual); Results first posted 2022-01-19 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: COVID-19; Sars-CoV-2
Keywords: rapid detection; assay; coronavirus; saliva
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Repeat Testing for SARS-CoV-2 (Experimental): Anyone over the age of 5yrs old with consent to provide a saliva sample for SARS-CoV-2 assay will be eligible to participate. Assay takes 20 minutes.
  Interventions: Device: Saliva Assay

INTERVENTIONS:
Device: Saliva Assay — saliva assay test for high concentrations of SARS-CoV-2

SUMMARY:
The purpose of this research study is to determine if high-frequency, rapid turn-around SARS-CoV-2 surveillance testing with this assay is feasible and able to be optimized to enable isolation and follow-up diagnostic testing. This test will be performed at various locations in the Madison, Wisconsin area using a mobile laboratory or standard lab space for processing. Saliva samples can be collected and processed at these locations or participants can self-collect at home and drop their samples off at designated locations for same day processing. Up to 10000 participants will be recruited for this study.

DETAILED DESCRIPTION:
Virtually all COVID-19 RNA assays require centralized laboratories. Samples collected in locations including public testing sites, workplaces, nursing homes, and residential housing are transported to centralized laboratories for testing, leading to lengthy delays in results reporting. The window of maximal contagiousness is thought to be only a few days, so these delays create the risk of excess transmission. Current testing methods are painful, which encourages testing hesitancy. Rapid, onsite detection of SARS-CoV- 2 RNA from non-invasive saliva could overcome these issues and provide a pathway to high throughput detection of people at the greatest risk of SARS-CoV-2 transmission but the logistics of such a testing program require real-world prototyping.

The purpose of this research study is to determine if high-frequency, rapid turn-around SARS-CoV-2 surveillance testing with this assay is feasible and able to be optimized to enable isolation and follow-up diagnostic testing. The investigators are also looking to see if it can be simplified so minimally trained staff can perform it successfully. The test is designed to identify people who are most contagious and likely to spread the virus to others. This test will be performed at various locations in the Madison area using a mobile laboratory or standard lab space for processing. Saliva samples can be collected and processed at these locations or participants can self-collect at home and drop their samples off at designated locations for same day processing. Results of potential findings of clinical significance will be communicated to the participants by a physician with appropriate expertise on the study team. Individuals with a potential finding of clinical significance will be encouraged to self-isolate and obtain a diagnostic test at their earliest convenience. No results will be given if the test is negative. If the participant consents, advanced molecular testing such as polymerase chain reaction (PCR) viral load tests, viral sequencing or other optimizing experiments can be done. Results of the viral sequencing can be shared via online databases, presentations and publications along with the date, site and county of collection to help facilitate tracking the spread of the virus. Study data will be shared via open research portals and online dashboards.

Participants with a potential finding of clinical significance will be contacted by phone approximately 1 week after the finding and asked the following questions. There will be 2 attempts at obtaining answers.

Question 1: Did you self-isolate after receiving the clinician's notification? Question 2: Did you receive a follow-up diagnostic test?

To assess whether or not the assay can be simplified so that minimally trained personnel can perform it, the investigators will perform proficiency tests with inactivated virus with newly trained staff which will help us optimize and refine the protocol. Successfully training staff achieve "proficiency" by correctly differentiating blinded positive and negative samples. This is how the investigators will assess the simplicity of the assay. For example, if a round of proficiency testing results in only 2/6 trainees achieving proficiency on their first try, that would suggest that the assay still has reducible complexity.

Tolerability of frequent testing could be done by keeping track of the interval between sample donations. Does the participant give a sample on a regular basis? Did they register but not donate a sample until weeks later? The study team will actively look for improved ways to assess this objective as we gather more data at these testing sites.

Relevant feasibility study is documented separately in NCT04460690.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide informed consent.
* Willing to provide informed consent and spit into a vessel (i.e cup or tube).
* Individuals at least 18 years old or between 5-17 years old and have a parent or legal guardian present to consent.
* Adult subjects must have decision-making capacity to provide consent on their own behalf.
* Participants must be able to speak English

Exclusion Criteria:

* Participants must not have visual or hearing impairments, or low literacy, that would prevent them from reading the consent form and interacting with a member of the research team to ask questions and receive responses during the consent process.
* Under 18 years of age with no parent or legal guardian present or under the age of 5 yrs
* Cannot speak English

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David O'Connor, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants will consent to having their data (not their name) and viral sequences shared with the public via manuscripts, presentations and online databases; the study team will share that with other researchers when needed. Samples can be shared with UW researchers internally and non UW researchers through the Material Transfer Agreement process.
Time Frame: Data from this study may be requested from other researchers 7 years after the completion of the primary endpoint by contacting David O'Connor at the University of Wisconsin -Madison.

REFERENCES:
- See also: Dave O'Connor's Lab — https://dho.pathology.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Repeat Testing for SARS-CoV-2
Started | 464
Number of Individuals Trained In COVID-19 Assay | 11
Completed | 464
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Repeat Testing for SARS-CoV-2
Number analyzed (Participants) | 464
Age, Customized [Count of Participants; unit: Participants] — Population: Participant age was not collected.
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Participant gender was not collected.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 464

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant Phone Surveys Conducted
Description: All participants with a potential finding of clinical significance (a result indicated the possible presences of SARS-CoV-2 in the saliva sample) will be contacted by phone approximately 1 week after the finding and asked if they received a follow-up diagnostic test and if they self-isolated after receiving the clinician's notification. There will be 2 attempts at obtaining answers. The investigators hope to receive at least 10 survey responses. This is a measure of surveillance feasibility.
Time Frame: up to 1 week after test
Population: 3 participants had a potential finding of clinical significance and were contacted.
Measure: Number; unit: phone surveys
Arm/Group | Repeat Testing for SARS-CoV-2
Number analyzed (Participants) | 3
phone surveys | 3

2. Primary Outcome: Number of Minimally Trained Personnel Who Achieve Assay Proficiency
Description: Successfully trained staff achieve "proficiency" by correctly differentiating blinded positive and negative samples. This is measure of the simplicity of the assay. Training personnel will take place over several months, proficiency should be determined within the same day as personnel are trained.
Time Frame: up to 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Repeat Testing for SARS-CoV-2
Number analyzed (Participants) | 11
Participants | 11

ADVERSE EVENTS:
Time Frame: Participants were not monitored for adverse events during sample collection.
Description: Participants were able to donate a saliva sample using two different methods. The first being a drop box with no interaction with the study team (saliva samples were collected off site) and the second being an in person saliva sample collection at designate dates and times. Participants were not monitored for adverse events during sample collection.
Groups:
- Repeat Testing for SARS-CoV-2: Participants were not monitored for adverse events during sample collection.
Arm/Group | Repeat Testing for SARS-CoV-2
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT04579549/Prot_SAP_002.pdf
  • Informed Consent Form (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT04579549/ICF_000.pdf